CLINICAL TRIAL: NCT06706427
Title: A Phase I/II Study for Subretinal Injection of NGGT001 in Patients With Bietti Crystalline Corneoretinal Dystrophy
Brief Title: Safety and Efficacy Study of NGGT001 in Bietti Crystalline Corneoretinal Dystrophy Subjects
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NGGT (Suzhou) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NGGT001-P-2301
Record Dates: First submitted 2024-11-14; First posted 2024-11-26 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Bietti Crystalline Corneoretinal Dystrophy
Keywords: BCD; Bietti Crystalline Corneoretinal Dystrophy
MeSH Terms: conditions — Bietti Crystalline Dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NGGT001 (Experimental): Single Arm: This study is a single-arm design in which all participants receive the NGGT001 gene therapy administered via subretinal injection. Participants are divided into three dose-escalation groups to evaluate safety and efficacy.
  Interventions: Biological: NGGT001

INTERVENTIONS:
Biological: NGGT001 — Using a recombinant adeno-associated virus (AAV) vector to deliver the gene CYP4V2 via subretinal injection for the treatment of crystalline retinal degeneration.

SUMMARY:
The objective of this study is to evaluate the safety, tolerability, and efficacy of subretinal injection of NGGT001 in patients with Bietti Crystalline Corneoretinal Dystrophy (BCD) and to recommend the optimal dosage for future clinical administration.

ELIGIBILITY:
1. Age ≥ 18 years old.
2. Male or female.
3. Confirmed diagnosis of BCD.
4. Molecular diagnosis confirmed cytochrome P450 family 4 subfamily v member 2 (CYP4V2) mutation.
5. AAV2 neutralizing antibody titer ≤1:5120.
6. 0.05 ≤ Best Corrected Visual Acuity (BCVA) ≤ 0.3.
7. -6.00D ≤ Refractive error ≤ +3.00D.
8. Agree to take contraceptive measures from the start of the study until one year after medication administration.
9. Volunteer to participate in the study and sign informed consent.

Exclusion Criteria:

1. There are choroidal neovascularization or other ocular diseases caused by BCD, which are considered to affect the operation or interfere with the interpretation of clinical endpoint.
2. Patients with evidence of neovascularization or suspected neovascularization, and the presence of tubular reflectivity in the neuroepithelial layer as shown by OCT.
3. Those who had used any of the treatment drugs within 6 months before enrollment, such as Lucentis, Avastin, Conbercept, Triamcinolone acetonide, etc. These may affect the experimental observation.
4. The treated eyes have undergone intraocular surgery, such as photodynamic therapy (PDT), vitrectomy, periocular vascular bypass surgery, etc., or need intraocular surgery in the process of clinical research, such as cataract surgery, retinal laser therapy, etc.
5. Have used or may use systemic drugs that may cause eye damage, such as psoralen, tamoxifen, etc.
6. Highly sensitive or allergic to ingredients in the test drug (with allergic history of two or more drugs or food).
7. Physical examination, vital signs, and laboratory examination (such as blood routine, urine routine, blood biochemistry, coagulation function, immunology examination, etc.) are abnormal and clinically significant, or the investigators believe that the abnormal indicators have clinical significance.
8. There are diseases or medical histories that may affect drug safety or in vivo processes, especially cardiovascular, liver, kidney, endocrine, digestive tract, lung, nerve, blood, tumor, immune or metabolic disorders considered by investigators to be of clinical significance.
9. Participated in clinical trials of other drugs or medical devices within three months before enrollment.
10. Female patients who are pregnant or lactating.
11. Any other conditions which lead the investigator to determine the participant is unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2029-09-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) from baseline to 52 weeks. | 52 weeks
  To evaluate the incidence and severity of AEs, including serious AEs (SAEs) of subretinal injection of NGGT001 in patients with BCD.
Evaluate the improvement in BCVA compared to baseline at Week 12, 26 and 52. | Week 12, Week 26 and Week 52
  To evaluate the BCVA in ETDRS test of subretinal injection of NGGT001 from baseline to W12, 26 and 52.

SECONDARY OUTCOMES:
Assessment of microperimetry changes in dB compared to baseline at Week 12, 26 and 52. | Week 12, Week 26 and Week 52
  Retinal sensitivity will be assessed using the MP-3 Type Microperimeter. This will be measured in dB (decibels), and the retinal sensitivity analysis will be conducted based on these readings.
Assessment of contrast sensitivity (CS) changes in dB compared to baseline at Week 12, 26 and 52. | Week 12, Week 26 and Week 52
  Changes in contrast sensitivity (CS) will be evaluated, and the measurements will be analyzed in decibels (dB).
Assessment of Optical Coherence Tomography (OCT) retinal thickness changes compared to baseline at Week 12, 26 and 52. | Week 12, Week 26 and Week 52
  Retinal thickness will be measured using Optical Coherence Tomography (OCT), and the outcome will be expressed in micrometers (µm).
Assessment of Multi-Luminance Mobility Test (MLMT) score changes compared to baseline at Week 12, 26 and 52. | Week 12, Week 26 and Week 52
  Multi-Luminance Mobility Test (MLMT) will assess subjects' daily life quality across different lighting conditions. The results will be categorized by the different light intensity levels, and the aggregate scores will be used to assess mobility performance

OTHER OUTCOMES:
Assessment of Static Visual Fields (SVF) changes compared to baseline at Week 12, 26 and 52. | Week 12, Week 26 and Week 52
  Static Visual Fields (SVF): Changes in visual field sensitivity will be evaluated at Weeks 12, 26 and 52, compared to baseline. The measurements will be expressed in light sensitivity units (dB).
Assessment of Fundus Autofluorescence (FAF) retinal structural changes compared to baseline at Week 12, 26 and 52. | Week 12, Week 26 and Week 52
  Retinal structural changes will be assessed at Week 12 and 26, compared to baseline. Fundus Autofluorescence (FAF) imaging will be used to evaluate the intensity of autofluorescence, and changes will be assessed using a dB threshold to measure variations over time in comparison to baseline.
Assessment of Quality of Life Questionnaire score changes compared to baseline at Week 12, 26 and 52. | Week 12, Week 26 and Week 52
  Quality of Life Questionnaire score will be measured at Week 12, 26 and 52, compared to baseline.
Assessment of MNRead Test changes compared to baseline at Week 12, 26 and 52. | Week 12, Week 26 and Week 52
  MNRead Test results will be evaluated at Week 12, 26 and 52, compared to baseline, assessing vision function.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Southwest Hospital/Southwest Eye Hospital, Third Military Medical University (Army Medical University), Chongqing, Chongqing Municipality
  - Xiamen Eye Center of Xiamen University, Xiamen, Fujian

IPD SHARING:
Plan to Share IPD: No